CLINICAL TRIAL: NCT03833804
Title: Data-driven Strategies for Substance Misuse Identification in Hospitalized Patients
Brief Title: Data-driven Identification for Substance Misuse
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Wisconsin, Madison (Other)
Collaborators: Rush University Medical Center (Other); National Institute on Drug Abuse (NIDA) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Sequential | Masking: None | Purpose: Screening
Other Study IDs: 2022-0983; A534285 (Other: UW Madison); SMPH/MEDICINE (Other: UW Madison); 1R01DA051464 (NIH)
Record Dates: First submitted 2019-02-06; First posted 2019-02-07 (Actual); Results first posted 2025-10-24 (Actual); Last update posted 2025-10-24 (Actual); Status verified 2025-10

CONDITIONS: Substance Use; Substance Abuse; Substance-Related Disorders
Keywords: natural language processing; machine learning; artificial intelligence; clinical decision support; unhealthy alcohol use; opioid use disorder; illicit drug use
MeSH Terms: conditions — Substance-Related Disorders; Opioid-Related Disorders

STUDY DESIGN:
Intervention Model Description: Quasi-experimental design as an interrupted time series
Masking Description: No masking as the manual screen is already part of usual care and the automated screen will become usual care in the post-period of the pre-post design.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- SMART-AI: NLP (natural language processing) pre-screen (Experimental): Automated processing of clinical notes collected during routine care in first 24 hours of hospital admission to identify individuals at-risk for substance misuse to receive standard-of-care full screening and assessment, brief intervention, or referral to treatment (SBIRT) intervention.
  Interventions: Other: Processing of clinical notes in the EHR data collected during routine care
- Usual Care (No Intervention): Data collected before the intervention began

INTERVENTIONS:
Other: Processing of clinical notes in the EHR data collected during routine care — Clinical notes collected in the first day of hospital admission during usual care as input to natural language processing and machine learning algorithm.
  Arms: SMART-AI: NLP (natural language processing) pre-screen

SUMMARY:
The investigators propose to develop an open-source, publicly available machine learning model that health systems could download and apply to their electronic health record data marts to screen for substance misuse in their patients. The investigators hypothesize that the natural language processing algorithm can provide a standardized and interoperable approach for an automated daily screen on all hospitalized patients and provide better implementation fidelity for screening, brief intervention, and referral to treatment.

DETAILED DESCRIPTION:
In 2016, nearly 30% hospital discharges in the United States (US) had a major diagnostic category for a substance-use related condition. Substance misuse ranks second among principal diagnoses for unplanned 7-day hospital readmission rates. Despite the availability of Screening, Brief Intervention, and Referral to Treatment (SBIRT) interventions, substance misuse is not part of the admission routine and only a minority of patients are screened for substance misuse in the hospital setting. This is particularly problematic, since among hospitalized inpatients, the prevalence of substance misuse is estimated to be as high as 25%, greater than either the general population or outpatient setting. Practical screening methods tailored for the hospital setting are needed.

In the advent of Meaningful Use in the electronic health record (EHR), efficiency for alcohol detection may be improved by leveraging data collected during usual care. Documentation of substance use is common and occurs in over 96% of provider admission notes, but their free text format renders them difficult to mine and analyze. Natural Language Processing (NLP) and machine learning are subfields of artificial intelligence (AI) that provide a solution to analyze text data in the EHR to identify substance misuse. Modern NLP has fused with machine learning, another sub-field of artificial intelligence focused on learning from data. In particular, the most powerful NLP methods rely on supervised learning, a type of machine learning that takes advantage of current reference standards to make predictions about unseen cases

In the earlier version of an NLP and machine learning tool, the investigators successfully used data from clinical notes collected in the first 24 hours of hospital admission to reach a sensitivity and specificity above 70% for identifying alcohol misuse. With nearly 36 million hospital admissions in 2016, a substance misuse classifier has potential to impact millions.

In this study, the aim is to prospectively implement a substance misuse classifier to examine its effectiveness against current practice of all hospitalized adult patients at a tertiary health system. The health system has a mature screening system to examine substance misuse classifier performance against current practice of questionnaire screening.

The hypothesis is that the substance misuse classifier may provide a standardized, interoperable, and accurate approach to screen hospitalized patients. Successful implementation of the classifier in hospitalized patients is a step towards an automated and comprehensive universal screening system for substance misuse.

ELIGIBILITY:
Inclusion Criteria:

* Ages 18 years old to 89 years old
* Inpatient status during hospitalization
* Length of stay greater than 24 hours

Exclusion Criteria:

* Cannot participate in the usual care SBIRT intervention
* Death or obtunded during first 24 hours of admission
* Discharged against medical advice
* Transferred from another acute care hospital
* Transferred to another acute care hospital

Ages: 18 Years to 89 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 64996 (Actual)
Dates: Start 2022-09-19 (Actual); Primary Completion 2024-09-19 (Actual); Study Completion 2024-09-19 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Rush University Medical Center, Chicago, Illinois, United States

IPD SHARING:
Plan to Share IPD: Yes
The patient data are protected health information and unavailable to public but the algorithm will be shared. The investigators will serialize our best models developed using either pickle (a Python native mechanism for object serialization) or joblib (https://pythonhosted.org/joblib/) and write software that will be capable of reloading them and making predictions. The software will be distributed via github.com or similar web-based software hosting service.
Supporting Information: Analytic Code
Time Frame: 12 months after completion of study and available for at least five years on github.com
URL: http://github.com

REFERENCES:
- [Result] Afshar M, Phillips A, Karnik N, Mueller J, To D, Gonzalez R, Price R, Cooper R, Joyce C, Dligach D. Natural language processing and machine learning to identify alcohol misuse from the electronic health record in trauma patients: development and internal validation. J Am Med Inform Assoc. 2019 Mar 1;26(3):254-261. doi: 10.1093/jamia/ocy166. PMID 30602031
- [Derived] Rojas JC, Joyce C, Markossian TW, Chaudhari V, McClintic MR, Castro F, Fairgrieve AJ, Dligach D, Oguss MK, Churpek MM, Nikolaides J, Afshar M. Clinical Implementation of an AI Algorithm for Substance Misuse Screening in Hospitalized Adults. medRxiv [Preprint]. 2025 Nov 19:2025.11.17.25340323. doi: 10.1101/2025.11.17.25340323. PMID 41332823
- [Derived] Joyce C, Markossian TW, Nikolaides J, Ramsey E, Thompson HM, Rojas JC, Sharma B, Dligach D, Oguss MK, Cooper RS, Afshar M. The Evaluation of a Clinical Decision Support Tool Using Natural Language Processing to Screen Hospitalized Adults for Unhealthy Substance Use: Protocol for a Quasi-Experimental Design. JMIR Res Protoc. 2022 Dec 19;11(12):e42971. doi: 10.2196/42971. PMID 36534461
- See also: login page but full code not finalized for publishing — https://github.com/

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: The comparison groups are pre-intervention and intervention. data from 31432 people were assessed prior to the intervention in 2022-2023 and data from 33564 people were assessed with the intervention from 2023-2024: data from 64996 people were assessed in total.
Groups:
- Usual Care: Before intervention
- NLP (Natural Language Processing) Pre-screen: Automated processing of clinical notes collected during routine care in first 24 hours of hospital admission to identify individuals at-risk for substance misuse to receive standard-of-care full screening and assessment, brief intervention, or referral to treatment (SBIRT) intervention.
  Processing of clinical notes in the EHR data collected during routine care: Clinical notes collected in the first day of hospital admission during usual care as input to natural language processing and machine learning algorithm.
Period: Usual Care Data Collection (2022-2023)
Arm/Group | Usual Care | NLP (Natural Language Processing) Pre-screen
Started | 31432 | 0
Completed | 31432 | 0
Not Completed | 0 | 0
Period: SMART-AI Data Collection (2023-2024)
Arm/Group | Usual Care | NLP (Natural Language Processing) Pre-screen
Started | 0 | 33564
Completed | 0 | 33564
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- NLP (Natural Language Processing) Pre-screen: SMART-AI: Automated processing of clinical notes collected during routine care in first 24 hours of hospital admission to identify individuals at-risk for substance misuse to receive standard-of-care full screening and assessment, brief intervention, or referral to treatment (SBIRT) intervention.
  Processing of clinical notes in the EHR data collected during routine care: Clinical notes collected in the first day of hospital admission during usual care as input to natural language processing and machine learning algorithm.
- Total: Total of all reporting groups
Arm/Group | Usual Care | NLP (Natural Language Processing) Pre-screen: SMART-AI | Total
Number analyzed (Participants) | 31432 | 33564 | 64996
Age, Continuous [Mean (Standard Deviation); unit: years] | 56 (19) | 56 (19) | 56 (19)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 18458 | 19421 | 37879
  Male | 12974 | 14143 | 27117
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  White | 10524 | 11097 | 21621
  Black | 11139 | 11650 | 22789
  Hispanic | 7363 | 8061 | 15424
  Asian | 1047 | 1064 | 2111
  Other | 1058 | 1318 | 2376
  Unknown | 301 | 374 | 675
Region of Enrollment [Number; unit: participants]
  United States | 31432 | 33564 | 64996
Patient Class [Count of Participants; unit: Participants]
  Inpatient | 24231 | 25992 | 50223
  Observation | 7201 | 7572 | 14773
Admission Type [Count of Participants; unit: Participants]
  Elective | 13753 | 14652 | 28405
  Emergency | 17679 | 18912 | 36591
Elixhauser Comorbidity [Mean (Standard Deviation); unit: comorbidities] — Population: Elixhauser Comorbidity was unknown for some participants.
  comorbidities
    number analyzed (Participants) | 30668 | 32672 | 63340
    (all) | 2.8 (4.8) | 2.9 (4.9) | 2.9 (4.8)
Length of Stay (LOS) [Mean (Standard Deviation); unit: days] | 5.1 (6.5) | 4.9 (6.4) | 5.0 (6.5)
Insurance [Count of Participants; unit: Participants]
  Medicaid | 8728 | 8714 | 17442
  Medicare | 13111 | 14364 | 27475
  Private | 7438 | 8038 | 15476
  Self Pay | 431 | 666 | 1097
  Other | 204 | 186 | 390
  Unknown | 1520 | 1596 | 3116
Discharge [Count of Participants; unit: Participants]
  Home | 21176 | 23335 | 44511
  Home / Home Health | 5739 | 5528 | 11267
  Skilled Nursing Facility / Rehab | 2760 | 2812 | 5572
  Long Term Acute Care | 165 | 171 | 336
  Other Transfer | 98 | 162 | 260
  AMA | 412 | 385 | 797
  Psych | 104 | 93 | 197
  Other / Unknown | 50 | 74 | 124
  Hospice / Expired | 928 | 1004 | 1932

OUTCOME MEASURES:

1. Primary Outcome: Proportion of Patients That Had a Universal Screen Positive and Received SBIRT (Screening, Brief Intervention, or Referral to Treatment)
Description: The primary outcome is the proportion of patients who received SBIRT after a positive universal screen for being at risk for substance misuse. The design is an interrupted time-series prospective observational study.
Time Frame: 24 months
Measure: Count of Participants; unit: Participants
Groups:
- SMART-AI: Automated processing of clinical notes collected during routine care in first 24 hours of hospital admission to identify individuals at-risk for substance misuse to receive standard-of-care full screening and assessment, brief intervention, or referral to treatment (SBIRT) intervention.
  Processing of clinical notes in the EHR data collected during routine care: Clinical notes collected in the first day of hospital admission during usual care as input to natural language processing and machine learning algorithm.
Arm/Group | Usual Care | SMART-AI
Number analyzed (Participants) | 31432 | 33564
Participants | 1189 | 1144
Statistical Analysis 1: Comparison: Usual Care vs SMART-AI; Test type: Non-Inferiority — The investigators conducted a noninferiority analysis using a prespecified margin of 0.5%. The noninferiority margin was selected based on expert input from addiction medicine clinicians and implementation scientists, who agreed that a 0.5% absolute difference in the composite intervention rate would be clinically acceptable given the workflow and scalability benefits of automation. The margin was chosen to reflect a reasonable balance between clinical impact and operational gain; p = 0.20, One-sided independent samples z-test; z-test = 0.86

2. Secondary Outcome: All-cause Re-hospitalizations Following 6-months From the Index Hospital Encounter
Description: We will compare healthcare utilization outcomes in all patients between pre- and post-periods controlling for all patient demographic and clinical characteristics.
Time Frame: 12 months enrollment with 6 months follow-up for rehospitalization
Measure: Count of Participants; unit: Participants
Arm/Group | Usual Care | SMART-AI
Number analyzed (Participants) | 31432 | 33564
Participants | 9584 | 10241

ADVERSE EVENTS:
Time Frame: No plan per protocol to collect adverse events data.
Description: Investigators did not plan per protocol to examine all-cause mortality outside of the discharge disposition (data reported in baseline characteristics), serious adverse events, or other adverse events. Adverse Events and Deaths were not collected.
Groups:
- Usual Care: data collected before study intervention
Arm/Group | Usual Care | SMART-AI: NLP (Natural Language Processing) Pre-screen
All-Cause Mortality (participants affected / at risk) | 0/0 | 0/0
Serious Adverse Events (participants affected / at risk) | 0/0 | 0/0
Other Adverse Events (participants affected / at risk) | 0/0 | 0/0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2022-04-01): https://cdn.clinicaltrials.gov/large-docs/04/NCT03833804/Prot_SAP_001.pdf